CLINICAL TRIAL: NCT05591001
Title: A Comparative Study of the Effect of Propofol Infusion Versus the Combination of Ketamine and Dexmedetomidine Infusion on the Amplitude of Motor Evoked Potential in Pediatrics Undergoing Tethered Spinal Cord Surgeries a Randomized, Double-blinded Controlled Study
Brief Title: Effects of Anesthetic Infusion on the Amplitude of Motor Evoked Potential in Pediatrics Undergoing Tethered Spinal Cord Surgeries
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amany Hassan Saleh, Associate professor of anesthesia ,surgical intensive care and pain management ,Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: N-83-2022
Record Dates: First submitted 2022-10-17; First posted 2022-10-21 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Tethered Cord
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Ketamine; Propofol

STUDY DESIGN:
Intervention Model Description: forty six Children undergoing untethered spinal cord surgery will be randomly allocated into two equal groups using computerized generated random tables.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: . The details of the series will be unknown to the investigators and the group assignment will be kept in a set of sealed envelopes, each bearing only the case number on the outside. a person who will prepare the drugs and data collector is not one of the trial investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine-dexmedetomidine group (Active Comparator): Dexmedetomidine( 0.4 -0.6 μg/.kg /.h r)) ketamine,( 1-2m/.kg/.hr) infusion and giving bolus of fentanyl,( 1-2μg/.kg/ ) with keeping mean arterial blood pressure and heart rates changes within 25% of the baseline.
  Interventions: Drug: ketamine and dexmeditomidine combination
- propofol group (Active Comparator): propofol (100 ug/kg/min) -giving a bolus of fentanyl, (1-2μg/.kg/ ) with keeping mean arterial blood pressure and heart rate changes within 25% of the baseline.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: ketamine and dexmeditomidine combination — Dexmedetomidine( 0.4 -0.6 μg/.kg /.hr)) ketamine,( 1 -2m/.kg/.hr) infusion
  Arms: Ketamine-dexmedetomidine group
Drug: Propofol — propofol (100 ug /kg/min) infusion
  Arms: propofol group

SUMMARY:
The tethered spinal cord is a common pathology in pediatric neurosurgery. Intraoperative neurophysiologic monitoring (IOM) has gained popularity over the past two decades as a clinical discipline that uses neurophysiologic techniques to detect and prevent iatrogenic neurologic injuries. IOM techniques are extensively used in adult neurosurgery and, in their principles, can be applied to the pediatric population. Inhalational agents cause a dose-dependent reduction in MEPs and are arguably considered incompatible with effective neurophysiological monitoring(5) For this reason, total intravenous anesthesia (TIVA), using IV anesthetics (propofol or ketamine) and opioids (fentanyl or remifentanil), is commonly used in spinal surgeries under MEPs monitoring

DETAILED DESCRIPTION:
A combination of ketamine and dexmeditomidine has several benefits in terms of hemodynamic stability, absence of respiratory depression, postoperative analgesia, and recovery. (11) ketamine could prevent the decrease of blood pressure and heart rate which had been observed with dexmedetomidine. In addition, dexmedetomidine could prevent the increase of blood pressure and heart rate, salivation, and physiological emergence reaction from ketamine. This combination was not previously used in this type of procedure except in a case report performed by Rozzana Penny who had used dexmedetomidine and ketamine infusion during scoliosis repair surgery with somatosensory and motor evoked potential monitoring in 15 years old female.(10) Evoked potentials are highly sensitive to fluctuations in physiological parameters such as peripheral and core body temperature, arterial blood pressure, hematocrit, etc. Keeping in view all the above factors we plan this study to compare the effect of the combinations of propofol and fentanyl versus the combination of ketamine and dexmedetomidine and fentanyl in producing a minimum effect on MEP amplitude and on hemodynamic stability during the surgery.

ELIGIBILITY:
Inclusion Criteria:

* children with ASA I and II presented to Abu elreesh hospital for untethered spinal cord surgery.

Exclusion Criteria:

* Children with neuromuscular diseases or congenital scoliosis.
* Children with growing rod distraction surgery.
* Children with American Society of Anaesthesiologists (ASA) physical status III, IV
* Children with preoperative use of antidepressant or anticonvulsant medications.
* Children with a known history of drug allergies.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
the mean microvolts of 3 measurements of MEPs at 5 minutes interval at AH muscle before skin incision. | 2 hours
  the amplitude of motor evoked potentials measures

SECONDARY OUTCOMES:
fentanyl consumption in micrograms | 2 hours
  total amount of fentanyl consumption intraoperatively
Measurement of MEP at baseline once the patient will be prone , at surgical incision , and once exposure of the spine will be complete and during spinal manipulation and At the end of the surgery. | 2 hours
  Microvolt of MEP at baseline
Measurements of blood pressure at base line T1, induction (T2) positioning( T3), skin incision (T4) , during spinal manipulation (T5)and by the end of the surgery (T6). | 2 hours
First rescue of analgesia | 2 hours
Side effects (sedation -hypotension ( MAP less than 25% from the baseline reading) - bradycardia - respiratory depression) | 6 hours
Measurements of heart rate at baseline T1, induction T2, positioning T3,spinal manipulationT4,at the end of surgery T5 | 2 hours
  Beats / minute?

CONTACTS AND LOCATIONS:
Locations (1):
- Amany Hassan Saleh, Giza, Egypt